CLINICAL TRIAL: NCT02199951
Title: Observational Study to Evaluate the Clinical Safety After Introduction of the Fixed Dose Artemisinin-based Combination Therapy Eurartesim® (Dihydroartemisinin/Piperaquine [Dha/Pqp]) in Public Health Districts in Sub-Saharan Africa.
Brief Title: Introduction of Eurartesim® in Burkina Faso, Mozambique, Ghana and Tanzania
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: INDEPTH Network (Other)
Collaborators: Ministry of Health, Ghana (Other Government); Ifakara Health Research and Development Centre (Other); Ministry of Health, Burkina Faso (Other Government); Centro de Investigacao em Saude de Manhica (Other)
Responsible Party: Sponsor
Other Study IDs: INESS 02/2012; GRANT ID#. 48363.01 (Other: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2013-05-01; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Malaria
Keywords: Uncomplicated Malaria; dihydroartemisinin; piperaquine
MeSH Terms: conditions — Malaria | interventions — artenimol; piperaquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dihydroartemisinin and piperaquine: The patients will take Eurartesim® (DHA/PQP) with a dose regimen of one administration every 24 hours over a period of three days, i.e. at Day 1, then after 24 hours (Day 2) and after 48 hours (Day 3) from the first administration. The dose will be based on body weight. Two strengths of Eurartesim® will be provided for dosing in children and adults: 20/160mg and 40/320mg of DHA and PQP respectively. Body weight (kg) Daily dose (mg) Number of tablets per dose 20/160mg DHA/PQ 40/320mg DHA/PQ 5 to <7 10 mg DHA and 80 mg PQP ½ tablet 7 to <13 20 mg DHA and 160 mg PQP 1 tablet 13 to < 24 40 mg DHA and 320 mg PQP 1 tablet 24 to < 36 80 mg DHA and 640 mg PQP 2 tablets 36 to < 75 120 mg DHA and 960 mg PQP 3 tablets 75 to < 100 160 mg DHA and 1280 mg PQP 4 tablets > 100.
  Interventions: Drug: Dihydroartemisinin and piperaquine

INTERVENTIONS:
Drug: Dihydroartemisinin and piperaquine — Antimalarial
  Other Names: Eurartesim

SUMMARY:
WHO recommends the use of artemisinin-based combination therapies (ACTs) in the treatment of uncomplicated malaria to stem falciparum malaria drug resistance. New ACTs are entering the African market and will be used by the public health care system. The collection of safety data and risk evaluation through observational data are critical in order to assess risk/benefit profile of each ACT through its life cycle and providing information on the best use. Additionally there is need to assess the impact of the introduction of a new ACT in the evolution of its efficacy and malaria morbidity and mortality. Dihydroartemisinin/Piperaquine (DHA/PQP) is a new ACT approved by European Medical Agency and a number of African countries. This is a phase IV observational evaluation of the clinical safety of the fixed-dose DHA/PQP (Eurartesim®) in public health facilities within selected Health and Demographic Surveillance Centres in Burkina Faso (Nouna), Mozambique (Manhica), Ghana (Dodowa, Kintampo, Navrongo), Tanzania (Rufiji) and other African countries to be added. Eurartesim® will be used as first-line treatment of uncomplicated malaria an objective to evaluate the safety of Eurartesim® when used under usual conditions in 10,000 patients. Patients > 6 months and 5 kg except pregnant women will be enrolled and Eurartesim® administered as a single daily dose regimen over 3 days. Patients will be contacted at Day 5 (± 2 days) after treatment, to assess recovery and any adverse events.

DETAILED DESCRIPTION:
Study will be performed in public health facilities in up to 7 selected HDSS centres (Health and Demographic Surveillance sites) within the HDSS in Burkina Faso (1), Mozambique (1), Ghana (3), and Tanzania (2), where Eurartesim® will be used as first-line treatment of uncomplicated malaria episodes.

Primary:

Evaluate the safety of Eurartesim® when used under usual conditions in 10,000 patients with signs and symptoms of uncomplicated malaria confirmed by a parasitological diagnosis (Microscopy/Rapid Diagnostic Test) or, when this test is not available, by WHO diagnostic criteria.

Main Secondary:

Intensive assessment of a nested subset of 1,000 patients to evaluate the effect of the administration of Eurartesim® on blood biochemistry, full blood count, WBC differential count and QTc intervals. QTc interval and piperaquine concentration relationship will also be investigated in selected centers.

Other Secondaries:

Although it is expected that the vast majority of patients will be infected with P. falciparum, comparisons of the clinical tolerability of Plasmodium falciparum infected patients versus patients infected with other Plasmodia, as confirmed by the thick blood smear results, will be carried-out in the nested subset of 1,000 patients.

Assessment of the relationship between the occurrence of Adverse Events and the administration of concomitant medications will also be evaluated in the subset of 1,000 patients.

All patients visiting Health facilities in the HDSS areas and for whom a diagnosis of uncomplicated malaria (according to the WHO criteria) is suspected or confirmed by a parasitological diagnosis (Microscopy/Rapid Diagnostic Test) and who have signed informed consent/assent (a parent/guardian for children below 18 years old) will be included in the study. In the subset of 1,000 patients, the presence of Plasmodia of any species will be confirmed microscopically.

A thick blood smear will be prepared for further microscopic diagnosis in all the patients. Eurartesim® tablets will be prescribed to the patients (or to the parents/guardians, if the patients are children) meeting the protocol inclusion criteria before the results of the thick blood smear are known.

The patients will be contacted at Day 5 (± 2 days), in order to capture recovery status and all the experienced adverse events. A visit by the community health agent will be scheduled on all the cases in which the information collected during the telephone contact should be considered incomplete or unreliable ones. Special procedures will be followed in case of serious and/or severe adverse events and events classified of special interest (see specific section).

The subset of 1,000 patients will be intensively followed-up. These patients will have haematology (Hb and full blood counts (RBC, WBC and differential count)) and standard biochemistry (BUN, Creatinine, ALT/AST, Bilirubine, electrolytes (K+ and Cl-)) undertaken at Day 1 (before drug administration), Day 3 (3-4 hours after the last dose of treatment), and Day 7. If the results are abnormal and clinically relevant, the blood examination will be repeated until normalization. In all the 1000 patients, a plasma sample will be collected on Day 1 (before drug administration), twice on Day 3 (i.e. before and 3-4 hours after the last drug administration) as well as on Day 7 to assess plasma PQ concentration. From such blood drawings and before centrifugation, three drops of whole blood will be spotted on filter papers. These filter papers will be utilized to determine whole blood piperaquine concentration with the Dry Blood Spot methodology (if a validated analytical method for such determination will be settled up at the time of the study course). ECGs will be undertaken on Day 1 (before drug administration), twice on Day 3 (i.e. before and 3-4 hours after the last drug administration) as well as on Day 7 (ECG on Day 1 and Day 3 after last drug administration will be collected in triplicate); safety information will be collected at all these visits.

If the QTcF (QT corrected by Fridericia's formula) value assessed on Day 3 before last dose is above 500 ms, Eurartesim® should be withheld until QTcF returns below 480 ms within 6 hours. Thereafter, the Eurartesim® cycle may be completed under frequent QTc monitoring based on medical judgment. If the QTcF does not return below 480 ms within 6 hours, another antimalarial therapy should be considered.

The occurrence of any adverse events will be solicited from the subset of 1,000 patients on Days 3 and 7 following administration of Eurartesim® as well as in any additional visits.

All patients in the study with a cardiac event of special interest (see below) will have an ECG performed.

Patients will be asked to report to the health facility or to the HDSS if any adverse event occurs after Day 5 (± 2 days) contact and within 28 days after the start of Eurartesim® intake.

Female patients will be encouraged to communicate to the study team if they get pregnant within a period of two months after the start of the Eurartesim® treatment. In these cases, information on the evolution of the pregnancy will be collected at 3, 6, 9 months and after the delivery (6 and 14 weeks). Information on the drugs taken during the pregnancy as well as AEs/SAEs/AESIs and the health status of the newborn/s will be collected.

Patients will be instructed to take Eurartesim® with a dose regimen of one administration every 24 hours over a period of three days, i.e. at Day 1, then after 24 hours (Day 2) and after 48 hours (Day 3) from the first administration.

The dose will be based on patient body weight. Two strengths of Eurartesim® will be provided to facilitate the dosing in children and adults: 20/160mg and 40/320mg of DHA and PQP respectively.

The patients will be instructed to take Eurartesim® with water, at least three hours before or three hours after food intake (i.e. three hours after the previous food intake with no food intake for the following three hours after Eurartesim® administration).

To facilitate drug administration in small children, tablets will be crushed on a spoon and given with water. If vomiting occurs within 30 min from drug administration, dose will be re-administered. If vomiting occurs within 30 to 60 min, half a dose have to be re-administered. Re-dosing should not be attempted more than once.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated malaria (Plasmodia of any species) diagnosed as per national policies and in line with WHO recommendations (a history of fever in the previous 24 h and/or the presence of anaemia, for which pallor of the palms appears to be the most reliable sign in young children). Confirmation of malaria by a parasitological diagnosis with RDT is encouraged but its absence does not prevent patients from being enrolled.

  * Age ≥ 6 months and weight ≥ 5 kg.
  * Capability of taking an oral medication.
  * Ability and willingness to participate based on signed informed consent (a parent or a guardian has to sign for children below 18 years old), or on verbal consent given in front of a witness signing the informed consent, and access to health facility. The patient is to comply with all scheduled follow-up visits.

Exclusion Criteria:

* • Known allergy to artemisinin or to piperaquine.

  * Known pregnancy.
  * Lactating women should be excluded if other anti-malarial treatments are available
  * Complicated malaria.
  * Taking medicinal products that are known to prolong the QTc interval. These include (but are not limited to):
  * Antiarrhythmics (e.g. amiodarone, disopyramide, dofetilide, ibutilide, procainamide, quinidine, hydroquinidine, sotalol).
  * Neuroleptics (e.g. phenothiazines, sertindole, sultopride, chlorpromazine, haloperidol, mesoridazine, pimozide, or thioridazine), antidepressive agents.
  * Certain antimicrobial agents, including agents of the following classes:
* macrolides (e.g. erythromycin, clarithromycin),
* fluoroquinolones (e.g. moxifloxacin, sparfloxacin),
* imidazole and triazole antifungal agents,
* and also pentamidine and saquinavir.

  * Certain non-sedating antihistamines (e.g. terfenadine, astemizole, mizolastine).
  * Cisapride, droperidol, domperidone, bepridil, diphemanil, probucol, levomethadyl, methadone, vinca alkaloids, arsenic trioxide.
  * Have taken a DHA/PQP dose in the previous four weeks.
  * Family history of sudden unexplained death, or personal or family history of predisposing cardiac conditions for arrhythmia/QT prolongation (including congenital long QT syndrome, arrhythmia, QTc interval greater than 450 milliseconds with either Bazett or Fridericia correction).

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with uncomplicated malaria except pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 28 Days
  • Clinical safety will be determined by analysis of the number of adverse events (frequency, intensity, action taken, outcome) captured during their follow up contacts on Day 5 (±2 days) after starting the treatment with Eurartesim® as well as those identified in the referring hospitals or through adverse events spontaneously reported by the patient detected at the health facility within 28 days after the first medication intake.

SECONDARY OUTCOMES:
Adverse events of special interest | 28 Days
  In case of an AESI confirmed by the study doctor, the sponsor shall be informed within 24 hours, even if the event does not satisfy any condition of seriousness. Notification will occur through the use of an ad hoc AESI form. AESIs can be related to:
  * Cardio-toxicity i.e. prolonged QT
  * Neurotoxicity/seizures
  * Cutaneous reactions/phototoxicity

OTHER OUTCOMES:
Peak plasma concentration (Cmax) on Day 3 and plasma concentrations before last dose on day 3 and day 7) | 7 Days
  In predefined centres having the capability to store plasma samples, all the 1000 subset will also perform a blood drawing for PQ plasma concentration at Day 1 (before drug administration), twice at Day 3 (before and 3-4 after the last drug administration) as well as on Day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Fred N Binka, MD, PhD, Principal Investigator — INDEPTH Network
Locations (7):
- Burkina Faso (2):
  - Nouna Research Centre, Nouna
  - Nanoro Health Research Centre, Ouagadougou
- Ghana (3):
  - INDEPTH Network, Accra
  - Dodowa Health ReseaRCH Centre, Accra
  - Kintampo Health Research Centre, Kintampo
- Mnahica Health Research Centre, Maputo, Mozambique
- Rufigi Research Centre, Rufiji, Tanzania

REFERENCES:
- [Derived] Wattanakul T, Ogutu B, Kabanywanyi AM, Asante KP, Oduro A, Adjei A, Sie A, Sevene E, Macete E, Compaore G, Valea I, Osei I, Winterberg M, Gyapong M, Adjuik M, Abdulla S, Owusu-Agyei S, White NJ, Day NPJ, Tinto H, Baiden R, Binka F, Tarning J. Pooled Multicenter Analysis of Cardiovascular Safety and Population Pharmacokinetic Properties of Piperaquine in African Patients with Uncomplicated Falciparum Malaria. Antimicrob Agents Chemother. 2020 Jun 23;64(7):e01848-19. doi: 10.1128/AAC.01848-19. Print 2020 Jun 23. PMID 32312783
- See also: INESS — http://www.indepth-network.org